CLINICAL TRIAL: NCT01283451
Title: Ability of Near Infrared Spectroscopy to Isolate Compartments of the Extremity
Status: Completed | Type: Observational
Sponsor: J&M Shuler (Industry)
Responsible Party: Sponsor
Other Study IDs: NIRS-01
Record Dates: First submitted 2011-01-24; First posted 2011-01-26 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Acute Compartment Syndrome
Keywords: near-infrared spectroscopy
MeSH Terms: interventions — Muscle Contraction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Exercise: NIRS values of all participants will be measured at baseline and following each 30-60 second exercise.
  Interventions: Behavioral: Muscle contraction

INTERVENTIONS:
Behavioral: Muscle contraction — Participants will perform a 30-60 second exercise designed to cause a temporary decrease in muscle oxygenation of a specific muscle group.

SUMMARY:
Near infrared spectroscopy (NIRS) provides a non-invasive means of continuously monitoring tissue oxygenation, which may be useful for diagnosis of acute compartment syndrome (ACS). Placement of these sensor pads on the surface of the skin must be such that light penetrates the intended compartment without inadvertently obtaining measurements of an adjacent compartment. The objective of this study is to examine whether the NIRS measurements of each compartment truly represent the tissue perfusion of the intended compartment, as indicated by the predictable decrease in muscle oxygenation of a given compartment in response to muscle fatigue. The investigators hypothesize that the tissue oxygenation values of the stimulated compartment will significantly decrease following muscle stimulation, indicating that the intended muscle compartment was successfully isolated. Additionally, the investigators hypothesize that NIRS values of unstimulated muscle compartments will not change from baseline.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* no current extremity injuries
* willing to provide written informed consent

Exclusion Criteria:

* history of any anatomy-altering surgery to the extremity in question
* history of peripheral vascular disease
* history of pulmonary disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study sample will consist of healthy volunteers recruited from the principle investigator's private practice.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Near infrared spectroscopy | <30 minutes
  NIRS values will be measured before and after muscle fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shuler, MD, Principal Investigator — Athens Orthopedic Clinic, PA
Locations (1):
- Athens Orthopedic Clinic, PA, Athens, Georgia, United States